CLINICAL TRIAL: NCT07374133
Title: Comparison of Intrathecal Morphine and Ultrasound-Guided Bilateral Transversalis Fascia Plane Block for Post-Cesarean Analgesia
Brief Title: Intrathecal Morphine vs Transversalis Fascia Plane Block After Cesarean Delivery
Status: Not yet recruiting | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilke Tamdogan, Asst.Prof.MD, Ondokuz Mayıs University
Other Study IDs: CS-TFPB
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Delivery; Postoperative Analgesia; Obstetric Anesthesia
Keywords: Cesarean Sections; Postoperative Pain; Analgesia; Ultrasonography, Interventional; Spinal Anesthesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective Cesarean Delivery Cohort: This cohort includes parturients aged 18-45 years undergoing elective cesarean delivery under spinal anesthesia. Participants are followed prospectively as a single cohort. Postoperative outcomes are compared between exposure groups defined by the routine clinical analgesic approach, including intrathecal morphine or ultrasound-guided bilateral transversalis fascia plane block.

SUMMARY:
This prospective single-center study compares intrathecal morphine and ultrasound-guided bilateral transversalis fascia plane block for postoperative analgesia in patients undergoing elective cesarean delivery under spinal anesthesia. The primary outcome is the number of parturients requiring rescue analgesia within the first 24 hours postoperatively. The secondary outcomes include postoperative pain scores, rescue analgesia requirement, nausea/vomiting, pruritus, and obstetric quality of recovery (ObsQoR-11T).

DETAILED DESCRIPTION:
This prospective single-center study investigates postoperative acute pain management in parturients aged 18-45 years undergoing elective cesarean delivery under spinal anesthesia.Participants will be followed as a single prospective cohort, and postoperative outcomes will be compared between exposure groups defined by the routine clinical analgesic approach (intrathecal morphine or ultrasound-guided bilateral transversalis fascia plane block).A total of 60 patients are planned to be enrolled. Eligible participants are term parturients with a gestational age greater than 37 weeks, classified as American Society of Anesthesiologists (ASA) physical status II, and scheduled for elective cesarean delivery under spinal anesthesia. Patients will be excluded if they refuse participation, undergo cesarean delivery under general anesthesia, have ASA physical status greater than III, multiple pregnancy, conversion to general anesthesia after spinal anesthesia, contraindications to central or peripheral regional anesthesia techniques, body mass index greater than 35 kg/m², known allergy or hypersensitivity to local anesthetics or opioids, or significant organ dysfunction such as severe hepatic or renal disease.

In routine clinical practice, the postoperative analgesic approach is determined through shared decision-making based on patient preference and the responsible anesthesiologist's clinical assessment. Accordingly, two postoperative analgesic strategies will be compared: addition of intrathecal morphine to spinal anesthesia and ultrasound-guided bilateral transversalis fascia plane block.

Following standard ASA monitoring, spinal anesthesia is performed in the sitting position at the L4-5 interspace using a 26-gauge spinal needle. After confirmation of free cerebrospinal fluid flow, 12.5 mg of 0.5% hyperbaric bupivacaine combined with 20 micrograms of fentanyl is administered intrathecally. In the intrathecal morphine group, 120 micrograms of morphine is added to the intrathecal anesthetic solution. Sensory block level is assessed using the pinprick test, and surgery is initiated when a T6 sensory level is achieved.

In the transversalis fascia plane block group, the block is performed in the postoperative period with the patient in the supine position. An ultrasound probe is placed transversely just cranial to the iliac crest, and the abdominal wall layers, transversalis fascia, retroperitoneal fat, and peritoneum are identified. Using an in-plane needle approach, after hydrodissection with 3 mL of normal saline, 20 mL of 0.25% bupivacaine is injected into the plane deep to the transversalis fascia. The procedure is repeated on the contralateral side.

For postoperative nausea and vomiting prophylaxis, 4 mg of intravenous ondansetron is administered near skin closure, and uterotonic agents are given according to institutional protocols. Postoperative analgesia consists of 1 g intravenous paracetamol every 8 hours and intramuscular diclofenac every 12 hours. When the Numeric Rating Scale (NRS) score exceeds 4, rescue analgesia is provided with 100 mg intravenous tramadol administered as a 30-minute infusion, with a maximum daily dose of 300 mg.

The primary outcome of the study is the number of participants requiring rescue analgesia within the first 24 hours postoperatively. Secondary outcomes include postoperative pain intensity assessed using the NRS at rest and during activity at 0, 3, 6, 12, and 24 hours; incidence and severity of postoperative nausea and vomiting assessed using a 0-4 verbal rating scale; incidence and severity of pruritus assessed using a 0-3 scale at the same time points; and patient satisfaction and quality of recovery assessed using the Obstetric Quality of Recovery-11T (ObsQoR-11T) questionnaire at 24 and 48 hours after surgery.

All data will be collected by an anesthesia resident not involved in the procedures, anonymized, and handled in accordance with the Declaration of Helsinki. The study will be reported in compliance with the STROBE reporting guidelines, and participant confidentiality will be strictly maintained.

ELIGIBILITY:
Inclusion Criteria:

* Female parturients aged 18 to 45 years
* Gestational age greater than 37 weeks
* American Society of Anesthesiologists (ASA) physical status II
* Scheduled for elective cesarean delivery under spinal anesthesia
* Willingness to participate in the study

Exclusion Criteria:

* Refusal to participate in the study
* Cesarean delivery performed under general anesthesia
* Conversion to general anesthesia after spinal anesthesia
* ASA physical status greater than III
* Multiple pregnancy
* Contraindications to central or peripheral regional anesthesia techniques
* Body mass index (BMI) greater than 35 kg/m²
* Known allergy or hypersensitivity to local anesthetics or opioids
* Presence of significant organ dysfunction (e.g., severe hepatic or renal disease)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of parturients aged 18-45 years undergoing elective cesarean delivery under spinal anesthesia at a single tertiary care center. Participants are followed prospectively as a single observational cohort, and postoperative outcomes are compared between exposure groups defined by the routine clinical analgesic approach, including intrathecal morphine or ultrasound-guided bilateral transversalis fascia plane block.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Requirement for Rescue Analgesia Within 24 Hours | Within the first 24 hours postoperatively
  The primary outcome is the number of participants who require rescue analgesia within the first 24 hours after cesarean delivery. Rescue analgesia is administered when the Numeric Rating Scale (NRS) pain score exceeds 4 and consists of intravenous tramadol given according to the institutional protocol.

SECONDARY OUTCOMES:
Postoperative Pain Intensity (NRS) at Rest | 0, 3, 6, 12, and 24 hours postoperatively
  Pain intensity at rest assessed using the Numeric Rating Scale (NRS, 0-10; higher scores indicate worse pain) at predefined postoperative time points.
Postoperative Pain Intensity (NRS) During Activity | 0, 3, 6, 12, and 24 hours postoperatively
  Pain intensity during activity assessed using the Numeric Rating Scale (NRS, 0-10; higher scores indicate worse pain) at predefined postoperative time points.
Postoperative Nausea and Vomiting (PONV) Severity Score | 0, 3, 6, 12, and 24 hours postoperatively
  Severity of postoperative nausea and vomiting assessed using a 0-4 verbal rating scale at predefined postoperative time points.
Pruritus Severity Score | 0, 3, 6, 12, and 24 hours postoperatively
  Severity of pruritus assessed using a 0-3 scale at predefined postoperative time points.
Obstetric Quality of Recovery (ObsQoR-11T) Total Score | 24 and 48 hours postoperatively
  Quality of recovery assessed using the Obstetric Quality of Recovery-11T (ObsQoR-11T) questionnaire. Total score range is 0-110, with higher scores indicating better recovery.

CONTACTS AND LOCATIONS:
Overall Officials: İlke TAMDOGAN, Study Director — Giresun University Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Serifsoy TE, Tulgar S, Selvi O, Senturk O, Ilter E, Peker BH, Ozer Z. Evaluation of ultrasound-guided transversalis fascia plane block for postoperative analgesia in cesarean section: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2020 Feb;59:56-60. doi: 10.1016/j.jclinane.2019.06.025. Epub 2019 Jun 27. PMID 31255890
- [Result] Jemal B, Mohammed F, Tesema HG, Ahmed S, Mohammed A, Regasa T, Obsa MS. Analgesic Efficacy of Spinal Morphine in Comparison With Transversus Abdominis Plane Block for Postoperative Pain Management in Patients Undergoing Cesarean Section Under Spinal Anesthesia: A Randomized Controlled Trial. Front Med (Lausanne). 2022 Feb 9;9:814538. doi: 10.3389/fmed.2022.814538. eCollection 2022. PMID 35223910
- [Result] Bilgin S, Aygun H, Genc C, Dost B, Tulgar S, Kaya C, Sertoz N, Koksal E. Comparison of ultrasound-guided transversalis fascia plane block and anterior quadratus lumborum block in patients undergoing caesarean delivery: a randomized study. BMC Anesthesiol. 2023 Jul 21;23(1):246. doi: 10.1186/s12871-023-02206-w. PMID 37480008